CLINICAL TRIAL: NCT06868381
Title: A Phase IIa, Single-Site, Open-Label Trial of Baricitinib in Patients With Cardiac Sarcoidosis
Brief Title: A Trial of Baricitinib in Patients With Cardiac Sarcoidosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Matthew C. Baker, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79204
Record Dates: First submitted 2025-03-03; First posted 2025-03-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Sarcoidosis
Keywords: baricitinib; sarcoidosis; cardiac sarcoidosis; Janus kinase inhibitor; JAK inhibitor
MeSH Terms: conditions — Sarcoidosis | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- baricitinib + steroid-sparing drug +/- glucocorticoid taper (Experimental): * Participants will be treated with baricitinib 4 mg daily for up to 16 weeks in combination with a background steroid sparing medication
  * Participants who are on steroids at the time of enrollment will continue the steroid at a dose of prednisone (or equivalent) ≤ 20mg PO daily at Baseline and complete an 8 week taper of their steroid medication per a standardized protocol
  Interventions: Drug: Baricitinib (LY3009104) 4 mg

INTERVENTIONS:
Drug: Baricitinib (LY3009104) 4 mg — baricitinib 4 mg tablet taken orally once daily

SUMMARY:
The goal of this clinical trial is to learn if baricitinib in combination with a background steroid-sparing medication can treat active cardiac sarcoidosis in adults. The main question it aims to answer is:

- In patients with active cardiac sarcoidosis, does treatment with baricitinib improve cardiac sarcoidosis disease activity as assessed by changes on cardiac FDG-PET/CT?

Participants will:

* Take baricitinib in combination with a steroid-sparing therapy for up to 16 weeks
* Visit the clinic every two to four weeks for checkups and tests
* Be asked to complete questionnaires to see how they feel on baricitinib and medication diaries to record when they take baricitinib

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of cardiac sarcoidosis based on one of the following pathways:

  * Histological Diagnosis

    * Myocardial or extracardiac biopsy demonstrating non-caseating granuloma with no alternative cause identified AND
    * Abnormal FDG uptake on cardiac PET-CT conducted within six weeks of Screening, in a pattern consistent with active cardiac sarcoidosis AND
    * Exclusion of other causes for cardiac manifestations
  * Clinical Diagnosis

    * One or more of the following is present:

      * Steroid +/- immunosuppressant responsive cardiomyopathy or heart block
      * Unexplained reduced LVEF (< 40%) and/or segmental wall motion abnormalities not related to coronary artery disease or another defined cause
      * Unexplained sustained (spontaneous or induced) VT
      * Mobitz type II 2nd degree heart block or 3rd degree heart block
      * CT chest and/or FDG PET-CT showing features consistent with pulmonary sarcoidosis and/or hilar lymphadenopathy AND
    * Abnormal FDG uptake on cardiac PET-CT conducted within 6 weeks of Screening, in a pattern consistent with active cardiac sarcoidosis AND
    * Exclusion of other causes for cardiac manifestations
* Active cardiac sarcoidosis based on abnormal FDG uptake on cardiac PET-CT conducted within six weeks of Screening, in a pattern consistent with active cardiac sarcoidosis
* No current treatment with immunosuppressive medications other than a steroid-sparing medication (including methotrexate, leflunomide, azathioprine, or mycophenolate mofetil), and/or prednisone (or equivalent) at a dose of ≤ 20mg daily at Baseline

Key Exclusion Criteria:

* Receipt of a non-biologic DMARD or immunosuppressive agent other than methotrexate, leflunomide, azathioprine, mycophenolate mofetil, hydroxychloroquine, or glucocorticoids within 28 days prior to screening
* Receipt of a bDMARD or tsDMARD, including non-depleting B-cell-directed therapy (eg, belimumab), T cell costimulatory blockade (eg, abatacept), TNF-alpha inhibition (eg, infliximab, adalimumab, etanercept, golimumab, certolizumab pegol), interleukin-6 inhibition (eg, tocilizumab, sarilumab), interleukin-1 inhibition (eg, anakinra), JAK inhibition (eg, tofacitinib, upadacitinib, baricitinib), or other biologic immunomodulatory agent within 28 days prior to screening
* Receipt of any biologic B cell-depleting therapy (eg, rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab) in the 6 months prior to screening; receipt of such a B cell-depleting agent in the period 6-12 months prior to screening is exclusionary unless B cell counts have returned to ≥ LLN
* History of venous thromboembolism (VTE) or an increased risk for VTE
* Current smoking
* Estimated glomerular filtration rate < 30 mL/min/1.73 m2 by Modification of Diet in Renal Disease Study (MDRD) equation
* Blood tests at screening that meet any of the following criteria:

  * Hemoglobin < 7.5 g/dL
  * Neutrophils < 1000/mm3
  * Absolute lymphocyte count < 500/mm3
  * Platelets < 100 x 109/L
* Subjects with the following abnormal liver function tests:

  * Aspartate aminotransferase (AST) > 2x ULN
  * Alanine aminotransferase (ALT) > 2x ULN
  * Total bilirubin (TBL) > 2x ULN unless AST, ALT, and hemoglobin are within central laboratory normal range and the patient has a known history of Gilbert syndrome
* Active, clinically significant infection at the time of Screening
* Active malignancy or history of malignancy that was active within the last 5 years, except as follows:

  * In situ carcinoma of the cervix following apparently curative therapy > 12 months prior to screening,
  * Cutaneous basal cell or squamous cell carcinoma following apparently curative therapy, or
  * Prostate cancer treated with radical prostatectomy or radiation therapy with curative intent > 3 years prior to screening and without known recurrence or current treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with resolution of cardiac FDG uptake on PET-CT | From baseline to end of treatment at 16 weeks
  Resolution of FDG uptake will be determined by the consensus of two blinded nuclear medicine radiologists, in accordance with current SNMMI and ASNC guidelines

SECONDARY OUTCOMES:
Percent change in FDG avidity (SUVmax) in the cardiac lesion with greatest FDG avidity on PET-CT | From baseline to 8 weeks and end of treatment at 16 weeks
Percent change in total cardiac metabolic activity on FDG PET-CT | From baseline to 8 weeks and end of treatment at 16 weeks
  Total cardiac metabolic activity is total lesion glycolysis within the heart
Proportion of patients with resolution of extracardiac FDG uptake on PET-CT | From baseline to 8 weeks and end of treatment at 16 weeks
Percent change in FDG avidity (SUVmax) in up to six extracardiac lesions on PET-CT | From baseline to 8 weeks and end of treatment at 16 weeks
Percent change in total extracardiac metabolic activity on FDG PET-CT | From baseline to 8 weeks and end of treatment at 16 weeks
  Total extracardiac metabolic activity is total lesion glycolysis of extracardiac disease
Proportion of patients with resolution of cardiac FDG uptake on PET-CT | From baseline to 8 weeks and end of follow-up at 28 weeks
Change in sarcoidosis disease activity assessment | From baseline to 8 weeks and end of treatment at 16 weeks
  Sarcoidosis disease activity assessed with King's Sarcoidosis Questionnaire. Total score range: 0 to 100, with 100 indicating the highest quality of life
Change in fatigue assessment | From baseline to 8 weeks and end of treatment at 16 weeks
  Fatigue assessed with FACIT-F. Total score range: 0-52, lower scores correspond with more fatigue
Change from Baseline in Physician Disease Activity Visual Analogue Scale (VAS) | From baseline to 8 weeks and end of treatment at 16 weeks
  Physician rates patient's disease on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state
Change from Baseline in Patient Disease Activity Visual Analogue Scale (VAS) | From baseline to 8 weeks and end of treatment at 16 weeks
  Patient rates their disease on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state
Changes in ACE laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Changes in high-sensitivity troponin I laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Changes in NT-proBNP laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Changes in total IgG laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Changes in ESR laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Changes in CRP laboratory assessment | From baseline to 8 weeks and end of treatment at 16 weeks
Number of participants with safety endpoints of interest | From screening to end of follow-up at 28 weeks
  Safety endpoints of interest include hospitalization for cardiac events, implantation of a left ventricular assist device (LVAD), cardiac transplantation, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Baker, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No